CLINICAL TRIAL: NCT03117218
Title: Quantitative Analysis of 3T Whole Heart Coronary Magnetic Resonance Angiogram Improves Detection of Functionally Significant Coronary Artery Disease
Brief Title: Correlation Between Quantitative Analysis of Coronary MRA and FFR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Yeonyee E Yoon, MD, Associate Professor, Seoul National University Bundang Hospital
Other Study IDs: B-1408/262-006
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Coronary Artery Disease; Magnetic Resonance Angiography; Fractional Flow Reserve
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Coronary MR angiography — Quantitative analysis of coronary MR angiogram

SUMMARY:
This study aims to evaluate whether quantitative analysis of coronary MR angiogram would improve the detection of functionally-significant coronary artery stenosis.

DETAILED DESCRIPTION:
Coronary MR angiography is performed with a 3.0-T imager with 32-channel coils. Qunatitative analysis of coronary MR angiogram is evaluated on the basis of the signal intensity (SI) profile along the vessel. Quantitative analysis of coronary MR angiogram (QCMRA) is calculated as [1 - (SImin/SIref)] x 100, where SImin is minimal SI and SIref is corresponding reference SI. Diagnostic performance of quantitative analysis of coronary MR angiogram for predicting functional significant coronary stenosis was evaluated by using fractional flow reserve (FFR) as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* 1 or more coronary stenoses in the major coronary artery with a vessel diameter ≥ 2mm on coronary MR angiogram
* Patient who were planned to undergo invasive coronary angiography and fractional flow reserve

Exclusion Criteria:

* clinically unstable patient
* a history of coronary revascularization
* infiltrative cardiomyopathy, hypertropic cardiomyopathy, myocarditis
* contraindication to use of adenosine
* complete occlusion of target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary stenosis on coronary MR angiograms who were planned to undergo invasive coronary angiography.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Estimated)
Dates: Start 2014-07-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-05-31 (Estimated)

PRIMARY OUTCOMES:
Presence of functionally significant coronary stenosis | within 1 month
  fractional flow reserve < 0.8

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hopsital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No